CLINICAL TRIAL: NCT01815775
Title: Predictive Value of Flow MRI in Normal Pressure Hydrocephalus Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI05-PR-LEGARS; 2006/0023 (Registry Identifier: DGS)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: Normal pressure hydrocephalus; flow MRI; dementia; cerebrospinal fluid; shunt
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Dementia | interventions — Hydrodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Normal pressure hydrocephalus (Experimental): Hydrocephalus patients planned for shunting surgery. They will undergo clinical and imaging examinations at day 1, 3 months and 1 year after their surgery.
  Interventions: Other: clinical and imaging examinations

INTERVENTIONS:
Other: clinical and imaging examinations — Quantitative CSF flow study was performed by 2D phase-contrast velocity-encoded cine MRI (repetition/echo time, 15/7 ms; field of view = 140 x 140 mm²; matrix size = 256 x 128, flip angle = 25 degrees,one excitation, slice thickness = 5 mm). Cerebrospinal fluid flow was measured with a velocity-encoding value of 10-20 cm/s. Peripheral gating was used to cover the entire cardiac cycle with retrospective cardiac synchronization of 32 quantitative flow-encoded images per cycle.
  Clinical examination consists in neuropsychological assessment (including mini mental state examination test and Bradley's scale) as well as Hakim's triad evaluation
  Other Names: flow MRI; cine phase-constrast magnetic resonance imaging; CSF pulsatility; hydrodynamic

SUMMARY:
The idea is to assess the predictive value of flow magnetic resonance imaging (flow MRI) for patient suffering normal pressure hydrocephalus (NPH) planned for surgery. By now, the depletive lumbar puncture is the best test assessing the efficacy of a forthcoming surgery. The idea is to demonstrate that flow MRI can be as effective as lumbar puncture in term of predictive value of surgery response.

In that way, cerebrospinal fluid (CSF) dynamics are evaluated by a single non invasive examination. CSF flow is measured at the Sylvius' aqueduct, cervical, arachnoid space and 4th ventricle levels.

ELIGIBILITY:
Inclusion Criteria:

* age: over 20 years
* diagnostic of normal pressure hydrocephalus
* ventricular dilation visible on radiological examination
* patients gave their written informed consent

Exclusion Criteria:

* age: less than 20 years
* MRI contra-indication
* pregnancy
* lumbar puncture within 48 hours before MRI
* cardiac arrhythmia
* cerebral/lacunar stroke

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
CSF stroke volume | Day 1
  Measurement of CSF stroke volume via flow MRI at the Sylvius' aqueduct level

SECONDARY OUTCOMES:
Hakim's triad evaluation | Day 1
  Assessment of the signs of normal pressure hydrocephalus
Hakim's triad evaluation | Day 90
  Assessment of the signs of normal pressure hydrocephalus (follow-up)
Hakim's triad evaluation | Day 365
  Assessment of the signs of normal pressure hydrocephalus (follow-up)
Neuropsychological test | Day 1
  classical neuropsychological assessment (including mini mental status evaluation)
Neuropsychological test | Day 90
  classical neuropsychological assessment (including mini mental status evaluation) (follow up)
Neuropsychological test | Day 365
  classical neuropsychological assessment (including mini mental status evaluation) (follow up)
CSF stroke volume | Day 60
  Measurement of CSF stroke volume by flow MRI at the Sylvius' aqueduct level (follow-up)
CSF stroke volume | Day 365
  Measurement of CSF stroke volume by flow MRI at the Sylvius' aqueduct level (follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, Picardie, France

REFERENCES:
- [Result] Mouton Paradot G, Baledent O, Sallioux G, Lehmann P, Gondry-Jouet C, Le Gars D. [Contribution of phase-contrast MRI to the management of patients with normal pressure hydrocephalus: Can it predict response to shunting?]. Neurochirurgie. 2010 Feb;56(1):50-4. doi: 10.1016/j.neuchi.2009.12.007. Epub 2010 Jan 25. French. PMID 20097391